CLINICAL TRIAL: NCT06887049
Title: ARISE: Achieving Routine Intervention and Screening for Emotional Health: Randomized Controlled Trial
Brief Title: Achieving Routine Intervention and Screening for Emotional Health
Acronym: ARISE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: University of California, San Francisco (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Midwest Clinicians' Network (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: IRB24-0622; R01DK133603-02 (NIH)
Record Dates: First submitted 2025-03-13; First posted 2025-03-20 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Type 2 Diabetes Mellitus (T2DM); Diabetes Distress
Keywords: diabetes distress screening
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARISE Learning Community Arm (Experimental): Community Health Centers will be given an in-depth training on the ARISE screening and intervention algorithm
  Interventions: Behavioral: ARISE Learning Community Diabetes Distress Screening and Intervention
- ARISE Enhanced Care (Other): Community Health Centers will be given a brief training on the 7A's model of diabetes distress screening and intervention
  Interventions: Behavioral: ARISE Enhanced Care brief training

INTERVENTIONS:
Behavioral: ARISE Learning Community Diabetes Distress Screening and Intervention — In-depth training for frontline community health center staff on ARISE algorithm to screen for degree of diabetes distress using T2-DDAS Core. If positive, screen for sources of diabetes distress using T2-DDAS Sources. Discuss results with patient and make any relevant referrals.
  Arms: ARISE Learning Community Arm
Behavioral: ARISE Enhanced Care brief training — Brief training on American Diabetes Association guidelines for screening for diabetes distress using the 7A's model
  Arms: ARISE Enhanced Care

SUMMARY:
The purpose of this project is to evaluate the effectiveness of diabetes distress screening and intervention on patients with type 2 diabetes mellitus (T2DM).

DETAILED DESCRIPTION:
Diabetes mellitus (DM) affects 30 million people in the U.S.1 The prevalence of diabetes is higher among Hispanics (12.5%) and African Americans (11.7%) compared to non-Hispanic whites (7.5%). Managing type 2 DM (T2DM) can be complex and burdensome; patients must modify their diet and exercise habits, take medications, check their blood sugars, visits their healthcare providers regularly, and navigate work and family life. Financial insecurity and social risks (e.g., transportation access) also disproportionately affect persons of color in the U.S. and in turn impede patients' ability to adhere to diabetes self-care recommendations. Diabetes distress (DD) is the stress, fear, and guilt in having to manage diabetes and is distinct from depression and anxiety. A meta-analysis of 58 international studies noted one in five adults with diabetes had elevated DD.6 DD has well documented associations with poor medication adherence, dietary and exercise behaviors, quality of life, and glycosylated hemoglobin (A1C). African-Americans and Hispanics have higher levels of DD compared to non-Hispanic whites.

The American Diabetes Association published guidelines promoting screening for and addressing DD as a critical part of clinical care. Multiple studies have tested standardized screening instruments for DD and intervention studies have demonstrated reductions in DD. However, only 24% of adults with diabetes report their health care team asked them how diabetes affected their lives and far fewer currently receive structured DD screening and follow-up. Efforts to systematically identify and address DD could be an important strategy to improve diabetes outcomes and address diabetes disparities. Community health centers (CHCs) can be important partners in this effort. CHCs provide primary care for 2.5 million adults with diabetes, of whom 30% have A1C >9% and 57% are racial ethnic minorities.

No studies have systematically implemented DD screening and treatment interventions into a real-world primary care setting or used a guideline based approach. To fill this gap, we developed the ARISE (Achieving Routine Intervention and Screening for Emotional health) intervention. ARISE is a primary care training and implementation program for clinicians and allied health professionals to support screening for and address DD in T2DM. ARISE utilizes a standardized process for screening adult patients with T2DM for DD using validated instruments, provides training and support for CHC staff applying evidence-based strategies on how to address DD in the encounter, and an algorithm for action steps and referrals based on individualized sources of DD (e.g. hypoglycemia, access based on social needs). This pragmatic study will compare ARISE to enhanced usual care (didactic lecture for clinical staff on emotional health of persons with diabetes) using a type I hybrid effectiveness-implementation design via a cluster randomized controlled trial. This study provides the opportunity to optimize T2DM care for populations with health disparities concordant with evidence-based guidelines to aid in the attainment of optimal glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* Patient at a participating clinic
* Type 2 diabetes
* Adult (18 years or older)
* A1C > 8%

Exclusion Criteria:

* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1250 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Rate of A1C across time | 12 months
  Rate of A1C from Baseline to follow-up

SECONDARY OUTCOMES:
Average diabetes distress score | 12 months
  Rate of diabetes distress at each community health center based on average of patients' "core" and "sources" screening scores (based on T2-DDAS screening)
Average of low density lipoproteins (LDL Cholesterol) measure | 12 months
  Rate of average measure of patients' cholesterol in the blood
Average systolic blood pressure across time | 12 months
  Average of patients' systolic blood pressure (measures the arterial pressure)
Average Body mass index at baseline and follow-up | 12 months
  Average of patients' BMI (a measure of height and weight)
Average depression screening (PHQ) | 12 months
  Average of patients' degree of depression based on survey
Average score of anxiety screening (GAD) | 12 months
  Average of patients' degree of anxiety based on survey
Average number of referrals across patients over time | 12 months
  Average of patients' number of referrals to other providers or resources, and frequencies of different types of referrals made (e.g., rate of patients sent to OBGYN, Ophthalmology, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Arshiya Baig, MD, MPH, Principal Investigator — University of Chicago; Danielle Hessler Jones, PhD, Principal Investigator — University of California, San Francisco

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fisher L, Polonsky WH, Hessler D. Addressing diabetes distress in clinical care: a practical guide. Diabet Med. 2019 Jul;36(7):803-812. doi: 10.1111/dme.13967. Epub 2019 May 7. PMID 30985025
- [Background] Chew BH, Vos RC, Metzendorf MI, Scholten RJ, Rutten GE. Psychological interventions for diabetes-related distress in adults with type 2 diabetes mellitus. Cochrane Database Syst Rev. 2017 Sep 27;9(9):CD011469. doi: 10.1002/14651858.CD011469.pub2. PMID 28954185
- [Background] Shin, P., Sharac, J., Barber, Z., Rosenbaum, S., & Paradise, J. (2015, March). Community Health Centers: A 2013 Profile and Prospects as ACA Implementation Proceeds. The Henry J. Kaiser Family Foundation. Retrieved from http://kff.org/medicaid/issue-brief/community-health-centers-a-2013-profileand-prospects-as-aca-implementation-proceeds/
- [Background] Health Resources and Services Administration (HRSA). Health Center Program. Table 7. Health Outcomes and Disparities. National Data. Available at: https://data.hrsa.gov/tools/datareporting/program-data/national/table?tableName=7&year=2020.
- [Background] Schmidt CB, van Loon BJP, Vergouwen ACM, Snoek FJ, Honig A. Systematic review and meta-analysis of psychological interventions in people with diabetes and elevated diabetes-distress. Diabet Med. 2018 Jun 13. doi: 10.1111/dme.13709. Online ahead of print. PMID 29896760
- [Background] Wagner H, Pizzimenti JJ, Daniel K, Pandya N, Hardigan PC. Eye on diabetes: a multidisciplinary patient education intervention. Diabetes Educ. 2008 Jan-Feb;34(1):84-9. doi: 10.1177/0145721707312205. PMID 18267994
- [Background] Nicolucci A, Kovacs Burns K, Holt RI, Comaschi M, Hermanns N, Ishii H, Kokoszka A, Pouwer F, Skovlund SE, Stuckey H, Tarkun I, Vallis M, Wens J, Peyrot M; DAWN2 Study Group. Diabetes Attitudes, Wishes and Needs second study (DAWN2): cross-national benchmarking of diabetes-related psychosocial outcomes for people with diabetes. Diabet Med. 2013 Jul;30(7):767-77. doi: 10.1111/dme.12245. PMID 23711019
- [Background] Fisher L, Hessler D, Glasgow RE, Arean PA, Masharani U, Naranjo D, Strycker LA. REDEEM: a pragmatic trial to reduce diabetes distress. Diabetes Care. 2013 Sep;36(9):2551-8. doi: 10.2337/dc12-2493. Epub 2013 Jun 4. PMID 23735726
- [Background] Polonsky WH, Fisher L, Earles J, Dudl RJ, Lees J, Mullan J, Jackson RA. Assessing psychosocial distress in diabetes: development of the diabetes distress scale. Diabetes Care. 2005 Mar;28(3):626-31. doi: 10.2337/diacare.28.3.626. PMID 15735199
- [Background] Welch GW, Jacobson AM, Polonsky WH. The Problem Areas in Diabetes Scale. An evaluation of its clinical utility. Diabetes Care. 1997 May;20(5):760-6. doi: 10.2337/diacare.20.5.760. PMID 9135939
- [Background] LeBron AM, Valerio MA, Kieffer E, Sinco B, Rosland AM, Hawkins J, Espitia N, Palmisano G, Spencer M. Everyday discrimination, diabetes-related distress, and depressive symptoms among African Americans and Latinos with diabetes. J Immigr Minor Health. 2014 Dec;16(6):1208-16. doi: 10.1007/s10903-013-9843-3. PMID 23689972
- [Background] Sturt J, Dennick K, Hessler D, Hunter BM, Oliver J, Fisher L. Effective interventions for reducing diabetes distress: systematic review and meta-analysis. International Diabetes Nursing. 2015;12(2):40-55.
- [Background] Skinner TC, Joensen L, Parkin T. Twenty-five years of diabetes distress research. Diabet Med. 2020 Mar;37(3):393-400. doi: 10.1111/dme.14157. Epub 2019 Oct 31. PMID 31638279
- [Background] Dennick K, Sturt J, Speight J. What is diabetes distress and how can we measure it? A narrative review and conceptual model. J Diabetes Complications. 2017 May;31(5):898-911. doi: 10.1016/j.jdiacomp.2016.12.018. Epub 2017 Feb 14. PMID 28274681
- [Background] Snoek FJ, Bremmer MA, Hermanns N. Constructs of depression and distress in diabetes: time for an appraisal. Lancet Diabetes Endocrinol. 2015 Jun;3(6):450-460. doi: 10.1016/S2213-8587(15)00135-7. Epub 2015 May 17. PMID 25995123
- [Background] Indelicato L, Dauriz M, Santi L, Bonora F, Negri C, Cacciatori V, Targher G, Trento M, Bonora E. Psychological distress, self-efficacy and glycemic control in type 2 diabetes. Nutr Metab Cardiovasc Dis. 2017 Apr;27(4):300-306. doi: 10.1016/j.numecd.2017.01.006. Epub 2017 Jan 31. PMID 28274728
- [Background] Dennick K, Sturt J, Hessler D, et al. High rates of elevated diabetes distress in research populations: A systematic review and meta-analysis. International Diabetes Nursing. 2015;12(3):93-107.
- [Background] Fisher L, Skaff MM, Mullan JT, Arean P, Mohr D, Masharani U, Glasgow R, Laurencin G. Clinical depression versus distress among patients with type 2 diabetes: not just a question of semantics. Diabetes Care. 2007 Mar;30(3):542-8. doi: 10.2337/dc06-1614. PMID 17327318
- [Background] Fisher L, Gonzalez JS, Polonsky WH. The confusing tale of depression and distress in patients with diabetes: a call for greater clarity and precision. Diabet Med. 2014 Jul;31(7):764-72. doi: 10.1111/dme.12428. PMID 24606397
- [Background] Walker RJ, Strom Williams J, Egede LE. Influence of Race, Ethnicity and Social Determinants of Health on Diabetes Outcomes. Am J Med Sci. 2016 Apr;351(4):366-73. doi: 10.1016/j.amjms.2016.01.008. PMID 27079342
- [Background] Hill-Briggs F, Adler NE, Berkowitz SA, Chin MH, Gary-Webb TL, Navas-Acien A, Thornton PL, Haire-Joshu D. Social Determinants of Health and Diabetes: A Scientific Review. Diabetes Care. 2020 Nov 2;44(1):258-79. doi: 10.2337/dci20-0053. Online ahead of print. No abstract available. PMID 33139407
- [Background] Centers for Disease Control and Prevention. National diabetes statistics report, 2020. Atlanta, GA: Centers for Disease Control and Prevention, US Department of Health and Human Services. 2020:12- 15.